CLINICAL TRIAL: NCT06742697
Title: Flexibility, Resistance, Aerobic, Movement Execution (FRAME) Training Program to Improve Gait Capacity in Adults With Hereditary Spastic Paraplegia: Protocol for a Single-cohort Feasibility Trial
Brief Title: Flexibility, Resistance, Aerobic, Movement Execution Training in Adults With Hereditary Spastic Paraplegia
Acronym: FRAME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1130
Record Dates: First submitted 2024-12-12; First posted 2024-12-19 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Hereditary Spastic Paraplegia
Keywords: feasibility; gait; endurance; speed; balance; neurorehabilitation; hereditary spastic paraplegia; motor learning; aerobic exercise; high intensity interval training; resistance training; flexibility training; gait training
MeSH Terms: conditions — Spastic Paraplegia, Hereditary | interventions — Pliability

STUDY DESIGN:
Intervention Model Description: Single-cohort feasibility trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HSP Cohort (Experimental): The whole cohort of HSP patients will receive the same comprehensive neurorehabilitation program aiming at improving gait capabilities (speed and endurance). The content and the dosis of the treatment will be personalized according to patient's specific needs and preferences.
  Interventions: Behavioral: Flexibility, Resistance, Aerobic, Movement Execution training

INTERVENTIONS:
Behavioral: Flexibility, Resistance, Aerobic, Movement Execution training — Flexibility: static and dynamic stretching combined with sensory, high-frequency electrical stimulation to reduce spasticity and improve mobility.
  Resistance training: core stability and lower limb strength training in conditions of instability, to improve strength, coordination, and balance.
  Movement execution training: gait training according to motor learning principles.
  Aerobic exercise: in the form of high-intensity interval training at the end of each session, to improve cardiovascular status and foster motor learning consolidation (probably due to the release of brain derived neurothrophic factors).

SUMMARY:
Hereditary Spastic Paraplegia (HSP) is a diverse group of genetic neurological conditions causing progressive weakness and spasticity in the lower limbs, severely reducing balance and gait capabilities. There is currently a lack of structured neurorehabilitation programs aimed at improving gait in adults with HSP. This protocol seeks to assess the feasibility and effectiveness of a structured training approach focusing on flexibility, muscle strength, motor control, balance, and aerobic capacity.

To this end, twenty adults diagnosed with HSP will engage in 10 to 16 sessions, each lasting 60 to 120 minutes, guided by a therapist once or twice a week, depending on individual preferences. At the end of the program, participants will receive a transfer package, including written instructions (a manual) and video tutorials, to encourage ongoing exercise at home. Assessments will occur before the intervention (T0), immediately after (T1), and three months later (T2). The primary outcomes will measure the feasibility of the program, including recruitment, retention, adherence, the absence of adverse events, and patient satisfaction. Secondary outcomes will focus on improvements in gait capabilities such as gait endurance and gait speed.

DETAILED DESCRIPTION:
INTRODUCTION:

Hereditary Spastic Paraplegia (HSP) is a heterogeneous group of inherited neurological disorders characterized by progressive weakness and spasticity in the lower limbs, which significantly impairs walking abilities (endurance and speed). Despite several specific interventions for particular deficits already having been studied, there is currently a lack of comprehensive and structured neurorehabilitation programs designed to improve walking function in these patients. Therefore, this protocol aims to explore the feasibility and effectiveness of a composite training approach focused on improving flexibility, muscle strength, motor control, balance, and aerobic capacity.

STUDY OBJECTIVES:

Primary endpoint: Feasibility of the study, assessed by the following:

Sufficient recruitment rate, with 20 patients enrolled within 24 months from the study's initiation.

Adequate adherence to the treatment plan, defined by the completion of at least 75% of the planned treatment sessions, with a minimum of 10 treatment sessions.

Sufficient patient retention, defined as at least 75% of enrolled patients completing the study with adequate treatment adherence.

Absence of serious adverse events related to patient participation in the study.

Patient satisfaction with the healthcare received during the study.

Secondary endpoint: Therapeutic efficacy of the study, assessed by:

Improvement in walking endurance (6-Minute Walk Test). Improvement in walking speed (10-Meter Walk Test).

Exploratory objectives:

Improvement in overall functional condition (Spastic Paraplegia Rating Scale and the Hereditary Spastic Paraplegia - Self Notion and Perception Questionnaire).

Improvement in passive joint range of motion in the lower limbs (goniometer). Improvement in lower limb muscle strength (5 Times Sit-to-Stand Test). Improvement in standing balance (Functional Reach Test and stabilometric platform).

STUDY DESIGN: Open-label, non-randomized, uncontrolled interventional study.

STUDY POPULATION: Hereditary Spastic Paraplegia patients

SAMPLE SIZE: 20 patients

ELIGIBILITY:

Inclusion criteria:

Adults diagnosed with Hereditary Spastic Paraplegia. Presence of any functional deficit in the lower limbs affecting walking, such as muscle weakness, hypertonia, or balance issues.

Ability to walk independently, without physical assistance from another person, defined by a Functional Ambulation Category score of 3 or higher.

Ability to understand simple instructions, comprehend the purpose of the study, willingness to participate, commitment to at least 10 treatment sessions, and suitability for signing the informed consent.

Exclusion criteria:

Use of botulinum toxin or surgery to treat lower limb hypertonia within six months prior to study enrollment.

Contraindications for moderate physical activity, including stretching exercises, muscle strengthening, and aerobic training.

Withdrawal Criteria:

Voluntary withdrawal by the patient. Occurrence of adverse events or health issues that prevent continuation of the treatment plan.

Patient Replacement:

Recruitment will continue until 20 subjects are enrolled. Any patients who withdraw from the study will not be replaced.

METHODS:

Twenty adults diagnosed with HSP will participate in 10 to 16 therapist-guided sessions, each lasting 60 or 120 minutes, occurring once or twice a week depending on individual choice and capabilities. At the conclusion of the study, participants will receive an information package (manual and video tutorials) to support long-term home exercise. Evaluations will take place at three time points: before the intervention (T0), immediately after the intervention (T1), and three months post-intervention (T2). The primary objectives will focus on assessing the study's feasibility (recruitment, retention, adherence, absence of adverse events, and patient satisfaction). Secondary outcomes will evaluate improvements in walking ability and specific contributing factors, such as reduced spasticity, increased muscle strength, and improved balance.

INTERVENTION:

FRAME training is composed of four key components:

Component 1: Flexibility. To decrease muscle tone and enhance mobility, the therapist will apply a combination of stretching exercises and electrical stimulation, targeting areas such as the triceps surae, adductors, rectus femoris, and hamstrings. Electrical stimulation will utilize biphasic, high-frequency sensory stimulation (100 Hertz, pulse width 200 µs, and intensity just below the motor threshold) for a duration of 30 minutes, combined with stretching activities.

Component 2: Resistance Training (and Balance). The resistance training will focus on strengthening muscles typically weakened in individuals with Hereditary Spastic Paraplegia (HSP), especially the proximal muscles of the hip and trunk. To promote muscle engagement and improve balance and coordination, core stability and resistance exercises will be performed under conditions of mild instability. These exercises will be carried out in sitting or standing positions, rather than lying down, to optimize muscle activation.

Component 3: Movement Execution (and Balance). Gait training will be based on motor learning principles such as repetitive, task-oriented practice, variable practice, and graded practice. Graded practice involves breaking down a complex movement into simpler segments, practicing each segment until proficiency is achieved, and then progressively combining them into more complex sequences. Patients will be challenged with standing balance exercises while working on specific gait impairments. Gait training will involve varying walking patterns, including fast, slow, sidewalk walking, walking backward, and stair climbing.

Component 4: Aerobic Training via High-Intensity Interval Training (HIIT). HIIT consists of brief, intense aerobic efforts using large muscle groups, followed by rest periods of equal length. HIIT has been found to produce better cardiovascular results with a lower perceived level of effort compared to moderate-intensity aerobic exercise. In this protocol, patients will perform 30-second high-intensity intervals followed by 30 seconds of passive rest, repeated 10 times in two sets. Each session will begin with a 5-minute warm-up, include a 5-minute rest between sets, and conclude with a 5-minute cool-down. Patients will participate in the modality most suitable for consistent training, such as walking, running, cycling, or squatting.

RELEVANCE:

This protocol is significant for providing clinicians with valuable insights into the feasibility and potential effectiveness of a comprehensive, clinically-oriented program designed to improve walking ability in adults with Hereditary Spastic Paraplegia. It also aims to inform future translational research studies in the field.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with Hereditary Spastic Paraplegia.
* Presence of any functional deficit in the lower limbs that affects walking, such as muscle weakness, hypertonia, or balance issues.
* Ability to walk without the need for physical contact with another person, as defined by a Functional Ambulation Category score of 3 or higher.
* Ability to understand simple instructions, comprehend the purpose of the study, willingness to participate and undergo at least 10 treatment sessions, eligible and willing to sign the informed consent.

Exclusion Criteria:

* Botulinum toxin or surgery to treat lower limb hypertonia in the six months prior to enrollment in the study.
* Contraindications for moderate physical activity, such as stretching exercises, muscle strength training, and aerobic capacity training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility (recruitment rate). | Enrolment (T0), end of treatment five to ten weeks after T0 (T1).
  Study feasibility in terms of achieving sufficient recruitment rate, defined as the enrollment of 20 patients within 24 months from the start of the study.
Feasibility (adherence rate). | Enrolment (T0), end of treatment five to ten weeks after T0 (T1).
  Study feasibility in terms of achieving adequate adherence to the treatment plan, defined as completing at least 75% of the scheduled treatment sessions, and in any case a minimum of 10 treatment sessions.
Feasibility (retention rate). | Enrolment (T0), end of treatment five to ten weeks after T0 (T1).
  Study feasibility in terms of achieving sufficient patient retention, defined as at least 75% of the enrolled patients completing the study with adequate adherence to the treatment.
Feasibility (safety). | Enrolment (T0), end of treatment five to ten weeks after T0 (T1).
  Study feasibility in terms of absence of any serious adverse event related to patient participation in the study.

SECONDARY OUTCOMES:
Six Minute Walking Test (6MWT). | Enrolment (T0), end of treatment five to ten weeks after T0 (T1), follow-up 12 weeks after T1 (T2).
  The 6MWT is a clinical assessment of gait endurance, by measuring the distance covered (metres) while walking on a straight even path (30 meters) for six minutes. According to original instructions, the patient is asked to walk along the path as fast as possible, taking turns at the edges of the path. Patients are allowed to walk autonomously or with assistive devices and to rest by standing.
Ten Metre Walk Test (10MWT). | Enrolment (T0), end of treatment five to ten weeks after T0 (T1), follow-up 12 weeks after T1 (T2).
  The 10MWT is used to assess walking speed in meters/second (m/s) over a short distance. The total time taken to walk six meters (the central portion of a 10-meter walkway) is recorded to the nearest hundredth of a second. 6 meters is then divided by the total time taken to ambulate and recorded in m/s.
  Two trials at comfortable pace are performed, followed by two trials at fast pace. Averages (one for comfortable pace, one for fast pace) are recorded.

OTHER OUTCOMES:
Passive range of motion. | Enrolment (T0), end of treatment five to ten weeks after T0 (T1), follow-up 12 weeks after T1 (T2).
  An inclinometer will be used to measure the passive range of motion for ankle dorsiflexion, knee flexion, hip abduction, and hip extension, on both sides.
Hereditary Spastic Paraplegia - Self Notion and Perception Questionnaire (HSP-SNAP). | Enrolment (T0), end of treatment five to ten weeks after T0 (T1), follow-up 12 weeks after T1 (T2).
  HSP-SNAP is a questionnaire used to assess the self-perception of individuals diagnosed with hereditary spastic paraplegia (HSP).
  HSP-SNAP includes 12 questions, with 2 items dedicated to each symptom dimension (stiffness, weakness, imbalance, reduced endurance, fatigue, and pain). Each pair of items for a given dimension includes both positive and negative responses to prevent automatic answers. The HSP-SNAP employs a 5-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree). To account for both positive and negative items, scoring is as follows: for items with a positive tone, the score is calculated as "patient's score minus 1" (pt score-1); for negative items, the score is "5 minus the patient's score" (5-pt score). The overall score is the sum of all item scores, ranging from 0 to 48. A higher score indicates better well-being and milder symptoms.
Functional Reach Test (FRT). | Enrolment (T0), end of treatment five to ten weeks after T0 (T1), follow-up 12 weeks after T1 (T2).
  FRT evaluates dynamic balance while standing. Patient is asked to stand with one shoulder flexed at 90 degrees and the hand making a fist, and then to bend forward up to the limit of balance, right before taking a step to prevent falling. A horizontal ruler taped on the wall is used to measure the difference in position of the head of the third metacarpal bone from starting to end position. Patients are not allowed to touch the wall or rotate the trunk while bending forward.
Five times Sit-to-Stand (5TSTS). | Enrolment (T0), end of treatment five to ten weeks after T0 (T1), follow-up 12 weeks after T1 (T2).
  The 5TSTS test is an assessment to evaluate lower body strength, balance, and functional mobility. The test involves the participant sitting in a chair, then standing up and sitting down five times as quickly as possible, without using their arms for assistance. The time taken to complete the five repetitions is recorded.
modified Spastic Paraplegia Rating Scale (mSPRS) | Enrolment (T0), end of treatment five to ten weeks after T0 (T1), follow-up 12 weeks after T1 (T2).
  The mSPRS is a clinical assessment tool used to evaluate the severity and progression of symptoms in individuals with hereditary spastic paraplegia. The scale measures aspects such as spasticity, mobility, and functional abilities related to walking, balance, and limb function.
  The mSPRS has a scoring range from 0 to 28, with higher scores on the mSPRS indicating more severe symptoms and greater impairment in motor function and spasticity.
Stabilometric platform. | Enrolment (T0), end of treatment five to ten weeks after T0 (T1), follow-up 12 weeks after T1 (T2).
  With the patient standing over a stabilometric platform, two kinematic assessments will be performed: (1) static stance, by standing for 30 seconds with eyes open and 30 seconds with eyes closed; (2) limits of stability, by bending with the body in different direction, displacing the centre of mass towards anterior, posterior, and lateral targets projected on a screen in front of the patient.
Isometric strength. | Enrolment (T0), end of treatment at four weeks (T1), follow-up at 12 weeks after T1 (T2).
  A dynamometer will be used to measure isometric strength for ankle dorsiflexors, ankle plantarflexors, knee extensors, knee flexors, hip extensors, hip flexors, hip abductors, on both sides.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Boccuni, PhD, Principal Investigator — Scientific Institute, IRCCS E. Medea, Department of Conegliano, Treviso, Italy.
Locations (2):
- Italy (2):
  - Scientific Institute, IRCCS E. Medea, Department of Bosisio Parini, Lecco, Italy., Bosisio Parini, Lombardy
  - Scientific Institute, IRCCS E. Medea, Department of Pieve di Soligo, Treviso, Italy, Pieve di Soligo, Veneto

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be shared with other researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start Date: June 2027. End Date: June 2037.
Access Criteria: Any researcher accredited by non-profit clinical and research centre.

REFERENCES:
- [Background] Eng JJ, Tang PF. Gait training strategies to optimize walking ability in people with stroke: a synthesis of the evidence. Expert Rev Neurother. 2007 Oct;7(10):1417-36. doi: 10.1586/14737175.7.10.1417. PMID 17939776
- [Background] Crozier J, Roig M, Eng JJ, MacKay-Lyons M, Fung J, Ploughman M, Bailey DM, Sweet SN, Giacomantonio N, Thiel A, Trivino M, Tang A. High-Intensity Interval Training After Stroke: An Opportunity to Promote Functional Recovery, Cardiovascular Health, and Neuroplasticity. Neurorehabil Neural Repair. 2018 Jun;32(6-7):543-556. doi: 10.1177/1545968318766663. Epub 2018 Apr 20. PMID 29676956
- [Background] Thijs L, Voets E, Denissen S, Mehrholz J, Elsner B, Lemmens R, Verheyden GS. Trunk training following stroke. Cochrane Database Syst Rev. 2023 Mar 2;3(3):CD013712. doi: 10.1002/14651858.CD013712.pub2. PMID 36864008
- [Background] Maccora S, Torrente A, Di Stefano V, Lupica A, Iacono S, Pilati L, Pignolo A, Brighina F. Non-pharmacological treatment of hereditary spastic paraplegia: a systematic review. Neurol Sci. 2024 Mar;45(3):963-976. doi: 10.1007/s10072-023-07200-1. Epub 2023 Nov 16. No abstract available. PMID 37968432
- [Background] Bellofatto M, De Michele G, Iovino A, Filla A, Santorelli FM. Management of Hereditary Spastic Paraplegia: A Systematic Review of the Literature. Front Neurol. 2019 Jan 22;10:3. doi: 10.3389/fneur.2019.00003. eCollection 2019. PMID 30723448
- [Background] Ruano L, Melo C, Silva MC, Coutinho P. The global epidemiology of hereditary ataxia and spastic paraplegia: a systematic review of prevalence studies. Neuroepidemiology. 2014;42(3):174-83. doi: 10.1159/000358801. Epub 2014 Mar 5. PMID 24603320
- [Derived] Boccuni L, Bortolini M, Stefan C, Dal Molin V, Dalla Valle G, Martinuzzi A. Flexibility, Resistance, Aerobic, Movement Execution (FRAME) training program to improve gait capacity in adults with Hereditary Spastic Paraplegia: protocol for a single-cohort feasibility trial. Front Neurol. 2025 Feb 18;16:1441512. doi: 10.3389/fneur.2025.1441512. eCollection 2025. PMID 40040914